CLINICAL TRIAL: NCT06263894
Title: The Effect of the Alexander Technique on Labor Pain and Anxiety: A Randomized Controlled Trial
Brief Title: Alexander Technique on Labor Pain and Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MarmaraU-Ebe-ZDY-01
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Labor Pain; Anxiety
Keywords: Anxiety; Alexander Technique; Midwifery; Labor Pain
MeSH Terms: conditions — Labor Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: One experimental group and one conventional (control) group
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to reduce selection bias in determining the experimental and control groups, a computer-assisted randomization program (https://www.randomizer.org) will be used for pregnant women who meet the inclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The application of the Alexander Technique to the women included in the experimental group will be created by providing body awareness by directing their current posture and movements in line with three principles. In this way, self-management of the birth process in primiparous women will be established. In order to develop the body awareness of the primiparous woman, the Alexander Technique will be applied with the training program created by the researcher in line with the three principles.
  Interventions: Other: Experimental group
- Conventional group (Other): The conventional (control group) will receive routine midwifery care during the birth process. Routine midwifery care includes follow-up of the pregnant woman and the baby and uninterrupted midwife support during the birth process.
  Interventions: Other: Experimental group

INTERVENTIONS:
Other: Experimental group — Alexander technique will be applied to the experimental group.

SUMMARY:
This study will examine the effect of the Alexander Technique on labor pain and anxiety during labor. This study is designed as a randomized controlled experimental study. The population of the study consists of primiparous pregnant women who applied to Istanbul Provincial Health Directorate Başakşehir Çam and Sakura City Hospital, D-Block Maternity Hospital between November 2023 and May 2024. In calculating the sample size, G*Power (3.1.9.6) program was used to calculate the sample size with an error of 0.05, effect level of 0.5, power of 95%, and the required sample size for 2 groups was calculated as 34 people for each group with a total of 68 people.

DETAILED DESCRIPTION:
Pain during childbirth has been described as the most severe pain women experience throughout their life course. Labor pain is a result of physiologic changes in the uterus. Pharmacologic and nonpharmacologic methods are used in the management of pain, which is a physiologic process. Nonpharmacological methods help women to feel comfortable in labor and contribute to women to have a positive birth experience by providing relaxation and reducing pain perception through cognitive, psychological and physical methods (Adil et al., 2020; Thompson et al. 2019). In addition, midwives who are with the woman during the birth process use non-pharmacological methods in an independent role in the management of labor pain, and this is also effective in alleviating the burden on current health expenditures. Alexander Technique appears as a non-pharmacologic method. In the literature, there is no study on the application of the Alexander Technique in the management of labor pain. It is assumed that the current posture and position to be provided with the Alexander Technique will be effective on pain and anxiety during the birth process. It is necessary to conduct studies on the use of the Alexander Technique in the birth process and evaluate the results.

This study will be the first study on the Alexander Technique to be applied to women in labor. The research to be conducted is planned as a randomized controlled experimental study. The population of the study consists of 68 primiparous pregnant women who applied to Istanbul Provincial Health Directorate Başakşehir Çam and Sakura City Hospital, D-Block Maternity Hospital between November 2023 and May 2024. Simple random sampling method will be used for the sample of the study. Pregnant women included in the study will be informed about the study and 'Informed Consent Form' and 'Voluntary Consent Form' will be filled. 'Personal Information Form', 'Visual Analog Scale (VAS)', 'Beck Anxiety Scale (BAS)' and 'Oxford Birth Anxiety Scale (OWLS)' will be applied to the pregnant women included in the experimental group. After the initial data is collected, the principles in the Alexander Technique will be applied when the woman's cervical dilatation is 0-4 cm. The duration of the application is approximately 15 minutes and the researcher will take an active role with the woman accompanied by a counselor during this period. The second application will be applied when the cervical dilatation is 5-7 cm and the third application will be applied when the cervical dilatation is 8-10 cm. 'Visual Analog Scale (VAS)' will be applied after each application. 'Visual Analog Scale (VAS)', 'Beck Anxiety Scale (BAS)' and 'Oxford Birth Anxiety Scale (OWLS)' will be applied at the 2nd hour after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study,
* Between the ages of 18-35,
* Primiparous and singleton pregnant,
* Women at term (between 37 and 41 weeks of gestation) will be included in the study.

Exclusion Criteria:

* Risky pregnancies,
* Women who become pregnant as a result of assisted reproductive techniques,
* Delivery by caesarean section,
* Wanting to leave without working,
* Women undergoing analgesia at any stage of the labor process will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-02 (Estimated)

PRIMARY OUTCOMES:
Decreasing labor pain | During labor, the first assessment will be performed when cervical dilatation is 0-4 cm, the second assessment when cervical dilatation is 5-7 cm and the third assessment when cervical dilatation is 8-10 cm.
  Alexander Technique applied in labor pain management has a decreasing effect on labor pain.
Decreasing anxiety | During labor, the first assessment will be performed when cervical dilatation is 0-4 cm, the second assessment when cervical dilatation is 5-7 cm and the third assessment when cervical dilatation is 8-10 cm.
  The Alexander Technique applied in labor pain management has a reducing effect on anxiety during labor.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanefeld N, Glover L, Jomeen J, Wadephul F. Women's experiences of using the Alexander Technique in the postpartum: '...in a way, it's just as beneficial as sleep'. Midwifery. 2021 Dec;103:103155. doi: 10.1016/j.midw.2021.103155. Epub 2021 Oct 1. PMID 34655836
- [Result] Kinsey, D., Glover, L., & Wadephul, F. (2021). How does the Alexander Technique lead to psychological and non-physical outcomes? A realist review. European Journal of Integrative Medicine, 46, 101371.
- [Result] Klein SD, Bayard C, Wolf U. The Alexander Technique and musicians: a systematic review of controlled trials. BMC Complement Altern Med. 2014 Oct 24;14:414. doi: 10.1186/1472-6882-14-414. PMID 25344325